CLINICAL TRIAL: NCT03685487
Title: Decolonization of Patients Carrying S. Aureus Before Cardiac Surgery: Study of the Risk Factors Associated With Failure
Acronym: STAdécol
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 18CH049; 2018-001505-90 (Other: ANSM)
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-10

CONDITIONS: Staphylococcus Aureus
Keywords: decolonization; mupirocin; cardiac surgery
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with failures of decolonization S. aureus: patients with failures of decolonization S. aureus in their nose
  Interventions: Procedure: decolonization; Other: compliance questionnaire

INTERVENTIONS:
Procedure: decolonization — current practice : V1 : consultation to the service : nasal sample for all 5 days before surgery : order sent with decolonization procedure : nasal mupirocin, shower and mouthwash V2 : admission to the service : nasal sample for all and urine sample for decolonized patients V3 : nasal sample for all
Other: compliance questionnaire — We asked if the patient has done the whole decolonization procedure

SUMMARY:
Staphylococcus aureus nasal carriage is a well-known risk factor for S. aureus surgical site infections (SSI). According to a recent study demonstrating 60% reduction risk of SSI due this bacterium after patients' screening and decolonization, recent French and WHO guidelines recommend in cardiac surgery the decolonization of nasal S. aureus carriers before surgery. In practice the decolonization procedures are not well-defined according notably to the duration and time of delivery before surgery and doses of topical antimicrobial drugs. The aim of the proposed study is to investigate the factors associated with failures of S. aureus decolonization: carriage state, compliance with treatment, S. aureus capacity of internalization in nasal epithelial cells, resistance to antimicrobial drugs used. This study will allow (i) to measure the frequency of patients with residual S. aureus carriage just before surgery, whatever they have been decolonized or not, (ii) to characterize the S. aureus nasal carriage state of patients before surgery, and (iii) to investigate the adding value of mupirocin dosage in the nose and urines of decolonized patients as a marker of compliance and efficacy of the decolonization process.

ELIGIBILITY:
Inclusion Criteria:

* Patient to benefit from cardiac surgery scheduled at Saint-Etienne University Hospital
* Surgery of first intention (no resumption)
* Patient affiliated or entitled to a social security scheme
* Patient agreeing to participate in the study and having signed the informed consent

Exclusion Criteria:

* Surgery in a context of infection
* Surgery in an emergency and semi-emergency context
* Protected major patient
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be offered to all major patient who needs cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
number of participants with failure of decolonization of nasal carriers of S. aureus | just before surgery
  These patients were screened positive for S. aureus in nasal swab culture collected during the preoperative consultation of cardiac surgery, who received a decolonization prescription and who are again detected positive in culture for S. aureus on the nasal collection performed on admission to the surgery department (just before surgery).

SECONDARY OUTCOMES:
Prevalence of nasal carriage of S. aureus just prior to cardiac surgery in all patients | before surgery
Prevalence of nasal carriage of S. aureus 3 months after cardiac surgery in all patients | 3 months
Correlation between nasal dosing of mupirocin and compliance | 3 months
Correlation between mupirocin urine metabolite assay associated with mupirocin nasal dosing and decolonization efficacy (failure or not). | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Florence GRATTARD, MD, Principal Investigator — CHU de Saint Etienne
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No